CLINICAL TRIAL: NCT05542654
Title: Foot Massage Applied to Hypertensive Pregnant Women Bakirkoy Doctor Sadi Konuk Training and Research Hospital
Brief Title: The Effect of Foot Massage on Blood Pressure and Anxiety Levels in Pregnants With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, ilayda sel, Research Assistant, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Bakirkoystatehospital
Record Dates: First submitted 2022-09-06; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Pre-Eclampsia; Gestational Hypertension; Chronic Hypertension With Pre-Eclampsia; Superimposed Pre-Eclampsia
Keywords: Gestational hypertension; preeclampsia; foot massage; blood pressure; anxiety
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Foot Massage — Pregnant women in the intervention group were given a foot massage for 15 minutes each, for a total of 30 minutes for three days, while the control group did not receive foot massage.

SUMMARY:
This research was conducted as a prospective, experimental and randomised controlled research to determine the effect of foot massage applied to pregnant women with hypertension on blood pressure and anxiety levels.

DETAILED DESCRIPTION:
The sample of the research a total of 80 pregnants, 40 interventions and 40 in the control groups, which were randomly selected from hypertension pregnant women who applied to Health Sciences University Istanbul Bakırköy Doctor Sadi Konuk Training and Research Hospital (BEAH). After the participants were given written and verbal information about the research, the intervention group received a foot massage for three days, 15 minutes on each foot, for a total of 30 minutes, while the control group did not receive foot massage. In the research; Participant Promotion Form which contains questions about general health appearances and socio-demographic, gynecological and obstetric story, Vital Finding Monitoring Form to save blood pressure, pulse and breathing numbers restrained before and after foot massage, State and Trade Anxiety Inventory (STAI) which evaluates the level of anxiety, was used.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years and over and diagnosed with hypertension during or before pregnancy were included in the study.

Exclusion Criteria:

* Pregnant women who could not communicate in Turkish were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2020-11-08 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Three days
  Hypertensive disorder is a systolic blood pressure of 140 mmHg and a diastolic blood pressure of 90 mmHg and above that occurs after the 20th week of pregnancy. In this respect, blood pressure measurement is extremely important in pregnant women. In this study, a total of 30 minutes of foot massage, 15 minutes on each foot, was applied to pregnant women with hypertension in the intervention group for three days, and blood pressure was measured at regular intervals. (Before the massage, 5 minutes after the massage, 15 minutes after the massage, 30 minutes after the massage, 90 minutes after the massage, 120 minutes after the massage) No intervention was applied to pregnant women with hypertension in the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırkoy Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ejindu A. The effects of foot and facial massage on sleep induction, blood pressure, pulse and respiratory rate: crossover pilot study. Complement Ther Clin Pract. 2007 Nov;13(4):266-75. doi: 10.1016/j.ctcp.2007.03.008. Epub 2007 May 8. PMID 17950182
- [Background] Corrigan L, O'Farrell A, Moran P, Daly D. Hypertension in pregnancy: Prevalence, risk factors and outcomes for women birthing in Ireland. Pregnancy Hypertens. 2021 Jun;24:1-6. doi: 10.1016/j.preghy.2021.02.005. Epub 2021 Feb 14. PMID 33618054